CLINICAL TRIAL: NCT06922019
Title: Exploring UK Ambulance Clinicians' Experiences of Attending Out of Hospital Cardiac Arrest (OHCA) Incidents Involving Children: A Mixed Methods Study
Brief Title: Ambulance Clinicians' Experiences of Attending OHCA in Children
Status: Not yet recruiting | Type: Observational
Sponsor: University of Warwick (Other)
Collaborators: London Ambulance Service NHS Trust (Other); Resuscitation Council UK (Unknown)
Responsible Party: Principal Investigator, Keith Couper, Associate Professor, University of Warwick
Other Study IDs: SOC.19/23-24; 344286 (Other: IRAS)
Record Dates: First submitted 2025-02-12; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Out of Hospital Cardiac Arrest
Keywords: out of hospital cardiac arrest; paediatric; children; ambulance; emergency medical service
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Out of hospital cardiac arrest patients: Data will be collected relating to approximately 600 patients aged <18 years who were treated for out of hospital cardiac arrest by one UK ambulance service between 2021 and 2024
- Survey participants: Approximately 1,500 ambulance clinicians employed by National Health Service (NHS) ambulance trusts across the UK who participate in an online survey.
- Interview participants (recent exposure): Approximately 12-15 ambulance clinicians with recent (<12 months) exposure to an out of hospital cardiac arrest incident involving a child, who will participate in a semi-structured interview.
- Interview participants (historic exposure): Approximately 3-4 ambulance clinicians with historic (>12 months) exposure to an out of hospital cardiac arrest incident involving a child, who will participate in a semi-structured interview.
- Focus group participants: Up to 18 advanced/critical care paramedics who will participate in focus group discussions.

SUMMARY:
This research will explore ambulance clinicians' experiences of attending out of hospital cardiac arrest (OHCA) incidents involving children.

OHCA occurs when the heart stops beating. This is a time critical emergency that requires immediate treatment to maximise the changes of survival. OHCA affecting children is rare, but when it happens it is vital that paramedics and other ambulance clinicians can respond and deliver high quality care.

Because OHCA in children is rare, ambulance clinicians attend these incidents infrequently. Some clinicians may only ever attend this type of incident once in their career. These incidents are technically challenging for ambulance clinicians, and highly stressful. Evidence from other setting suggests that clinicians may be ill-prepared to manage these events.

This research aims to understand how OHCA incidents involving children are currently managed, and to explore the views and experiences of ambulance clinicians with respect to attending OHCA incidents involving children.

By learning from what is currently being done, and from clinicians' experiences, the research team aims to develop recommendations for how the response to these patients, and the support provided to ambulance clinicians, could be improved.

The research team will review the records of patients under the age of 18 who have been treated for OHCA by one ambulance service over a four-year period. Data will be collected from these records to allow the care delivered to be compared to international guidelines, and to explore what factors might influence the delivery of this care.

The research will also involve a survey of ambulance clinicians working across the UK to understand their experiences, and how prepared they feel to attend these incidents. Finally, the research team will undertake interviews with clinicians who have been involved in the management of a child with OHCA and focus group discussions with specialist clinicians to allow us to learn from their experiences.

DETAILED DESCRIPTION:
Work Package 1:

This work package comprises of a retrospective cohort study of patients under the age of 18 who have been treated for out of hospital cardiac arrest by one UK ambulance service.

Pseudonymised data will be collated for each patient included in the study, describing all actions taken by the ambulance service from the point the call for emergency help was received by the ambulance service to the time death was confirmed, or the patient was handed over to a receiving hospital team. These data will be collected in case report forms within a secure electronic database system.

Data will be extracted from electronic records (including computer aided dispatch and electronic patient care records) held by the ambulance service. A researcher based in the ambulance service will review each record to ensure complete data capture, supplementing the records with additional information not captured by the electronic data extraction as required (e.g. data entered into free text boxes or captured in handwritten records).

Descriptive statistics will be used to describe the management of patients included in the cohort, and to compare the management to UK and international guidelines. Further analysis will explore if patient management differs in the presence of certain patient, clinician, system, or situational factors.

Work Package 2:

The research team will conduct an online survey of ambulance clinicians working across UK ambulance services. The survey will be distributed through ambulance service sites across the UK and through social media.

Questions will include Likert-style and open questions to assess clinician attitudes and views in relation to their preparedness to respond to cardiac arrests in children. Questions will also explore previous experience of attending these incidents.

Recognising that clinicians involved in the resuscitation of a child may be at risk of psychological injury, respondents who report previous exposure to OHCA incidents involving children will be administered the validated 'Impact of Event Scale - Revised' (IES-R) questionnaire as part of the survey. IES-R is a 22-question instrument designed to measure symptoms of post-traumatic stress disorder (PTSD) in reference to a specific traumatic event. All participants who have attended OHCA incidents involving an adult will be administered IES-R with reference to the most recent event which will provide a comparator group to quantify if differences in the response to adult and child OHCA exist

Work Package 3:

Semi-structured interviews will be undertaken with 12-15 clinicians who have recently (in the previous 12 months) attended a child with out of hospital cardiac arrest (recent exposure interview cohort). In these semi-structured interviews, the research team will explore the clinicians experience during and following the incident, their perceived preparedness for attending the incident and their experiences of post-event support. A topic-guide will be developed for the interview which will include an opportunity to explore any emergent issues or concepts from the analysis of the clinician survey (WP2).

In addition, a small number of interviews (3-4) will be undertaken with clinicians who attended an out of hospital cardiac arrest incident involving a child earlier in their career (>12 months ago; historic exposure interview cohort). These interviews will follow the same format but will explore how perceptions and experiences of these events may have changed over time.

The research team will arrange 2-3 focus group discussions with specialist critical care ambulance clinicians (up to 6 clinicians per focus group; specialist clinician focus group cohort). These clinicians have a higher rate of exposure to out of hospital cardiac arrest incidents involving children, and by the nature of their dispatch models tend to arrive on scene later once interventions have been started. They will therefore have a unique insight into how their colleagues react to these incidents and the concerns expressed by these colleagues at the time or immediately following an incident.

The aim of these focus group discussions will be to explore this cadre of clinicians' experience of attending these events which may span many years and include a significant number of different events. Topic guides will be developed which will be influenced by the emerging themes from the clinician interviews. Where focus group discussions prove difficult to arrange, individual semi-structured interviews will be undertaken with eligible clinicians using the same topic guides.

ELIGIBILITY:
Out of hospital cardiac arrest patients

Inclusion Criteria:

* Patients attended by London Ambulance Service NHS Trust (LAS)
* Incidents occurring between January 2021 and December 2024
* Out of Hospital Cardiac Arrest recognised by LAS clinicians
* Aged under 18 years at the time the incident occurred

Exclusion Criteria:

* New born patients who had not taken their first spontaneous breath before cardiac arrest was recognised
* Incidents occurring outside of LAS' operational area (Greater London, UK)
* Patients who have registered an NHS National Data Opt-Out

Survey participants

Inclusion Criteria:

* Ambulance clinician (including registered healthcare professionals and non-registered ambulance clinicians)
* Currently responds to 999 calls (face to face) as part of their role
* Would be expected to attend a paediatric OHCA incident as part of their role
* Consents to participate in study

Exclusion Criteria:

* Non-clinical ambulance service employee
* Not employed by an NHS Ambulance Service in the UK

Interview participants (recent exposure)

Inclusion Criteria:

* Ambulance clinician (including registered healthcare professionals and non-registered ambulance clinicians)
* Employed by a participating NHS Ambulance Service Site
* Attended an out of hospital cardiac arrest incident involving a child (>1 day old, < 18 years old) in the 12 months prior to the proposed interview date
* Consents to participation in the study

Exclusion Criteria:

* Previously participated in an interview or focus group discussion as part of this study
* Employed in a specialist critical care role (e.g. Critical Care Paramedic)
* Attended an out of hospital cardiac arrest incident involving a child (>1 day old, <18 years old) within two weeks of the proposed interview date

Interview participants (historic exposure)

Inclusion Criteria:

* Ambulance clinician (including registered healthcare professionals and non-registered ambulance clinicians)
* Employed by a participating NHS Ambulance Service Site
* Attended an out of hospital cardiac arrest incident involving a child (>1 day old, < 18 years old) more than 12 months prior to the proposed interview date
* Consents to participation in the study

Exclusion Criteria:

* Previously participated in an interview or focus group discussion as part of this study
* Attended an out of hospital cardiac arrest incident involving a child (>1 day old, < 18 years old) within 12 months of the proposed interview date
* Employed in a specialist critical care role (e.g. Critical Care Paramedic)

Focus group participants

Inclusion Criteria:

* Ambulance clinician employed in a specialist critical care role (e.g. Critical Care Paramedic)
* Employed by a participating NHS Ambulance Service Site
* Consents to participation in the study

Exclusion Criteria:

* Previously participated in an interview or focus group discussion as part of this study
* Has not attended an out of hospital cardiac arrest incident involving a child (>1 day old, <18 years old) whilst working in a specialist critical care role (e.g. Critical Care Paramedic)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The out of hospital cardiac arrest patient group will include patients aged <18 years who were treated for out of hospital cardiac arrest by the London Ambulance Service NHS Trust.
  The survey, interview and focus group participants will be made up of ambulance clinicians employed in an NHS ambulance trust in the UK.
  * Survey participants in the recent exposure group will have recently attended an out of hospital cardiac arrest involving a child
  * Survey participants in the historic exposure group will have attended an out of hospital cardiac arrest involving a child >12 months before the interview date
  * Focus group participants will be specialist critical care paramedics who attend out of hospital cardiac arrest incidents involving children
Sampling Method: Non-Probability Sample
Enrollment: 2137 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Delivery of treatment in compliance with European Resuscitation Council Guidelines (work package one) | During cardiac arrest event (until handover at hospital or termination of resuscitation)
  Proportion of cases that receive treatment that complies with European Paediatric Advanced Life Support guidelines.
Preparedness of clinicians to attend OHCA involving children (work package two) | Baseline (defined as the date of survey completion)
  Measured using self-reported Likert scale
Clinician experiences of attending OHCA incidents involving children (work package three) | Baseline (defined as the date of interview/focus group participation)
  Measured through inductive thematic analysis of interviews and focus groups - data from interviews and focus groups will be combined and analysed thematically as one dataset to describe the overall experience of ambulance clinicians.

SECONDARY OUTCOMES:
Proportion of participants with moderate or high levels of symptoms consistent with PTSD following attending an OHCA incident involving a child (work package two) | Baseline (defined as the date of survey completion)
  Post Traumatic Stress Disorder (PTSD) symptoms will be measured using the The Impact of Event Scale - Revised (IES-R) with reference to an attended OHCA incident involving a child. Participants will be classified as having moderate or high levels of symptoms consistent with PTSD if their mean score across all questions is 2 or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Warwick, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No